CLINICAL TRIAL: NCT01963377
Title: Evaluation of Feasibility of Dedicated Extra O2-channel in a Bronchoscope.
Brief Title: Toward the Development of a Bronchoscope With a Dedicated O2 Channel ?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Vincent Ninane, Head of Department Pulmonology, Centre Hospitalier Universitaire Saint Pierre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: B076201215478; AK/12-11-90/4190 (Other: Comité d'éthique Saint Pierre)
Record Dates: First submitted 2013-10-09; First posted 2013-10-16 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Bronchoscopy; O2-supplementation
Keywords: bronchoscopy; O2-supplementation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Nasal Cannulae / 2. Bronchoscope channel (Experimental): Supplementation of O2 through will take place first through the aspiration channel of the bronchoscope, in second phase of the study O2-supplementation will be done through nasal cannulae.
  Interventions: Device: O2 through nasal cannulae; Device: O2-channel
- 1. Bronchoscope channel / 2. Nasal Cannulae (Experimental): Supplementation of O2 through will take place first through nasal cannulae, in second phase of the study O2-supplementation will be done through the aspiration channel of the bronchoscope.
  Interventions: Device: O2 through nasal cannulae; Device: O2-channel

INTERVENTIONS:
Device: O2 through nasal cannulae — supplementation of O2 through nasal cannulae during bronchoscopy
Device: O2-channel — supplementation of O2 through aspiration channel of bronchoscope during bronchoscopy

SUMMARY:
Feasibility of using an extra bronchoscopic channel for supplementation of oxygen will be studied by comparing O2-supplementation by nasal cannulae versus O2-supplementation through aspiration channel of the bronchoscope.

DETAILED DESCRIPTION:
Comparison of O2 administration using bronchoscope versus nasal cannulae in normal volunteers.

This study will compare partial pressure of oxygen measured in capillary blood (PcO2) at various O2 flow from 0 to 2 and 4 l/min administered using nasal cannulae or bronchoscope. During bronchoscopy, oxygen will be administered throughout the aspirating channel of the scope which extremity will be positioned at mid-tracheal level. After local anesthesia of the airways using lignocaine spray 10% and solution 1%, the bronchoscope will be introduced in seated position using a mouthpiece and placed at mid-tracheal level. Arterial O2-pressure sampled at the earlobe will be measured after incremental O2-supplementation from 0 to 2 and then 4 l/min using a nasal cannula or the aspirating channel of the bronchoscope. At each flow rate, capillary O2-pressure will be measured after 2 minutes. Between each condition of O2-supplementation there will be a pause of 5 minutes of room air breathing. The order of O2-supplementation condition will be selected at random. The whole bronchoscopic procedure should then last about 15 minutes. Additional doses of lignocaine 1% will be instilled in the trachea as requested and O2 saturation and heart rhythm will be monitored continuously during the procedure. Since the subjects are probably able to perceive additional flows in the nose and/or trachea and this may affect the pattern of breathing and the results, air at similar flow rate will be added in the nasal cannulae when O2 is administered using the bronchoscope channel and vice versa such that the subject will be blinded to the way O2 is administered.

This study should allow to demonstrate higher values of capillary O2-pressure during bronchoscopic administration of O2 than when using nasal cannulae. As shown by a recent meta-analysis, partial pressure of O2 measured in capillary blood from the arterialized earlobe (PcO2) is lower than the arterial value but this factor is not important in the present study since it will concentrate on differences in PO2 between the two conditions at similar O2 flow rates that are not affected by this limitation.

ELIGIBILITY:
Inclusion Criteria:

* healthy subject

Exclusion Criteria:

* younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
PcO2 difference | 1 hour
  PcO2 difference after different modes of O2-supplementation (nasal cannulae vs O2 through aspiration channel of bronchoscope) will be measured and compared

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ninane, Prof., MD, Principal Investigator — CHU St. Pierre
Locations (1):
- CHU St. Pierre, Brussels, BHG, Belgium